CLINICAL TRIAL: NCT00707694
Title: Searching for Longevity Genes in the Historically Unique Ashkenazi Jewish Population
Brief Title: The Longevity Genes in Founder Populations Project
Status: Recruiting | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH); American Federation for Aging Research (Other); Weill Medical College of Cornell University (Other); Boston University (Other); Regeneron Pharmaceuticals (Industry); Harvard Medical School (HMS and HSDM) (Other); Stanford University (Other); Tufts Medical Center (Other); Columbia University (Other); University of Minnesota (Other); Rutgers Health (Unknown); University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: 1998-125; 2U19AG056278-07A1 (NIH); 3U19AG056278-06S1 (NIH); P01AG021654 (NIH); 1R56AG088624-01 (NIH); R01AG088659 (NIH); G42988 (Other Grant/Funding Number: American Federation for Aging Research)
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Extreme Longevity
Keywords: 95 years of age and older

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Probands: Ashkenazi Jews ages 95 and older
- Offspring: Ashkenazi Jewish offspring of Ashkenazi Jewish parent(s) who lived to at least the age of 95
- Controls: Ashkenazi Jewish people with no family history of longevity

SUMMARY:
We believe extreme longevity is due to specific genes which function to delay aging and prevent disease. The purpose of the research is to identify the genes/mutations associated with healthier aging; to understand the biological functions of these genes/mutations; and to develop therapies to replicate these preservative genetic activities in individuals who do not have the genetic profile for longevity.

ELIGIBILITY:
Inclusion Criteria:

* Ashkenazi Jewish, age 95+,
* Offspring of person age 95+,
* Offspring of parents who died age 70 or younger.

Exclusion Criteria:

* Non-Ashkenazis

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Ashkenazi Jews:
  Ages 95 and older, their offspring and control group with no family history of longevity.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 1998-07 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nir Barzilai, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Private Homes, New York, New York
  - Hebrew Home Riverdale, Riverdale, New York

REFERENCES:
- [Result] DeVito LM, Barzilai N, Cuervo AM, Niedernhofer LJ, Milman S, Levine M, Promislow D, Ferrucci L, Kuchel GA, Mannick J, Justice J, Gonzales MM, Kirkland JL, Cohen P, Campisi J. Extending human healthspan and longevity: a symposium report. Ann N Y Acad Sci. 2022 Jan;1507(1):70-83. doi: 10.1111/nyas.14681. Epub 2021 Sep 8. PMID 34498278
- [Result] Moqri M, Herzog C, Poganik JR; Biomarkers of Aging Consortium; Justice J, Belsky DW, Higgins-Chen A, Moskalev A, Fuellen G, Cohen AA, Bautmans I, Widschwendter M, Ding J, Fleming A, Mannick J, Han JJ, Zhavoronkov A, Barzilai N, Kaeberlein M, Cummings S, Kennedy BK, Ferrucci L, Horvath S, Verdin E, Maier AB, Snyder MP, Sebastiano V, Gladyshev VN. Biomarkers of aging for the identification and evaluation of longevity interventions. Cell. 2023 Aug 31;186(18):3758-3775. doi: 10.1016/j.cell.2023.08.003. PMID 37657418
- [Result] Moqri M, Herzog C, Poganik JR, Ying K, Justice JN, Belsky DW, Higgins-Chen AT, Chen BH, Cohen AA, Fuellen G, Hagg S, Marioni RE, Widschwendter M, Fortney K, Fedichev PO, Zhavoronkov A, Barzilai N, Lasky-Su J, Kiel DP, Kennedy BK, Cummings S, Slagboom PE, Verdin E, Maier AB, Sebastiano V, Snyder MP, Gladyshev VN, Horvath S, Ferrucci L. Validation of biomarkers of aging. Nat Med. 2024 Feb;30(2):360-372. doi: 10.1038/s41591-023-02784-9. Epub 2024 Feb 14. PMID 38355974
- [Result] Bae H, Song Z, Ali A, Sasaki T, Tesi N, Lords H, Leshchyk A, Abe Y, Hirose N, Arai Y, Barzilai N, Weiss EF, Hulsman M, van der Lee S, van Schoor NM, Huisman M, Pijnenburg Y, van der Flier W, Reinders M, Holstege H, Milman S, Perls TT, Andersen SL, Sebastiani P. Increased genetic protection against Alzheimer's disease in centenarians. Geroscience. 2025 Jul 4. doi: 10.1007/s11357-025-01774-8. Online ahead of print. PMID 40615639
- [Result] Ali A, Zhang ZD, Gao T, Aleksic S, Gavathiotis E, Barzilai N, Milman S. Identification of functional rare coding variants in IGF-1 gene in humans with exceptional longevity. Sci Rep. 2025 Mar 25;15(1):10199. doi: 10.1038/s41598-025-94094-y. PMID 40133344
- [Result] Ying K, Castro JP, Shindyapina AV, Tyshkovskiy A, Moqri M, Goeminne LJE, Milman S, Zhang ZD, Barzilai N, Gladyshev VN. Depletion of loss-of-function germline mutations in centenarians reveals longevity genes. Nat Commun. 2024 Oct 19;15(1):9030. doi: 10.1038/s41467-024-52967-2. PMID 39424787
- [Derived] Barzilai N, Gabriely I, Atzmon G, Suh Y, Rothenberg D, Bergman A. Genetic studies reveal the role of the endocrine and metabolic systems in aging. J Clin Endocrinol Metab. 2010 Oct;95(10):4493-500. doi: 10.1210/jc.2010-0859. PMID 20926537